CLINICAL TRIAL: NCT05843175
Title: Maternal ExeRcIse Timing to Optimise Postprandial Glucose in Type 1 Diabetes
Acronym: MERIT1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Graz (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11954
Record Dates: First submitted 2023-03-27; First posted 2023-05-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy in Diabetic; Type 1 Diabetes
MeSH Terms: conditions — Pregnancy in Diabetics; Diabetes Mellitus, Type 1 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised, single-centre, controlled crossover in parallel groups (pregnant and non-pregnant women with type 1 diabetes)
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant women with type 1 diabetes (Experimental): Participants will undergo 3 experimental conditions in random order at week of gestation 16 and 35 (experimental phases 1 and 2): pre-meal exercise, post-meal exercise, and non-exercise meal.
  Interventions: Other: Exercise and meal testing (acute stimuli)
- Non-pregnant women with type 1 diabetes (Experimental): Participants will undergo 3 experimental conditions in random order after recruitment (experimental phase 1): pre-meal exercise, post-meal exercise, and non-exercise meal.
  Interventions: Other: Exercise and meal testing (acute stimuli)

INTERVENTIONS:
Other: Exercise and meal testing (acute stimuli) — Pre-meal exercise: 1º milkshake intake + 2º exercise test
  Post-meal exercise: 1º exercise test + 2º milkshake intake
  Non-exercise meal: Only milkshake intake

SUMMARY:
Poor glycaemic control in pregnancy is a major factor leading to obstetric complications and future maternal-offspring diseases. This phenomenon is evidenced in women with type 1 diabetes (T1DM), and is worrisome since it is aggravating the disease burden of this and next generations.

Exercise is a promising tool to improve glucose control during pregnancy and thus avoid adverse consequences.

The MERIT1D study will explore when is exercise (before or after lunch) more effective to improve postprandial glycaemic control in pregnant and non-pregnant women (of reproductive age) with T1DM, and the mechanisms underlying these metabolic responses.

DETAILED DESCRIPTION:
Poor glycaemic control in pregnancy is a major factor leading to obstetric complications and future maternal-offspring diseases (e.g., macrosomia, diabetes). This phenomenon is evidenced in women with type 1 diabetes (T1DM), and is worrisome since it is aggravating the disease burden of this and next generations. Therefore, to find strategies aimed at breaking this intergenerational cycle has become a high-priority. Exercise is a promising tool to improve short-term glycaemic responses such as postprandial glucose peaks and glucose variability, and thus reduce adverse maternal-neonatal outcomes. However, it is unknown which timing of exercise is more effective to optimise postprandial glycaemic control in pregnant women with T1DM, and non-pregnant women (of reproductive age) with T1DM. The mechanisms underlying these benefits in T1DM and pregnancy are also to be established.

The MERIT1D project will unravel which timing of exercise (before or after a meal at lunchtime) is more effective to optimise postprandial glycaemic control in pregnant and non-pregnant women with T1DM, and the mechanisms underlying these metabolic responses. Ten pregnant women with T1DM and ten non-pregnant women with T1DM will be involved in this randomised controlled crossover trial.

Pregnant women at gestational week 16 and 35 (experimental phases 1 and 2, respectively), and non-pregnant peers once after recruitment (experimental phase 1), will undergo 3 experimental conditions within 10 days (random order): pre-meal exercise, post-meal exercise, and non-exercise meal.

Each experimental phase will entail participants attending 4 times to the research centre. Therefore, pregnant women will come to the research centre for a total of 8 study visits, while non-pregnant women will come only to 4 study visits. The acute exercise stimulus will consist of a well-controlled submaximal walking test. The standardised meal provided will consist of a mixed milkshake equivalent to the 35 % of their resting energy expenditure, being made up of approximately 45% carbohydrates, 35% fat, and 20% proteins. Postprandial glycaemic responses will be continuously monitored using last-generation glucose monitoring systems during the 10-day period. Immunometabolic markers (e.g., lipids, cytokines) will be determined in maternal blood and placenta samples.

The MERIT1D study will contribute to the understanding of exercise timing in T1DM and pregnancy, and its underlying mechanisms. This will translate into a better clinical prediction, diagnosis, prognosis and treatment of glycaemic dysregulations, and into more effective exercise programmes for pregnant and non-pregnant women with T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women and non-pregnant women with T1DM aged 20-40 years
* Having a BMI of 18-29.9 kg/m2 at pre-pregnancy (pregnant women) or recruitment (non-pregnant)
* Clinical diagnosis of T1DM, or/and multiple daily insulin injections for >1 year, and/or using insulin pump therapy (open-loop).
* Willingness to provide informed consent to participate in the MERIT1D study.
* Being able to read and speak German, English or Spanish well enough to completely understand the instructions, provide informed consent and conduct the experimental procedures.

Exclusion Criteria:

* Having poor glycaemic control HbA1c>10% (86 mmol/mol).
* Recurrent severe hypoglycaemia; hospitalisation for diabetic ketoacidosis during the last year.
* Women who smoke or drink alcohol frequently, or require complex diets.
* Having polycystic ovarian syndrome, poorly controlled asthma/allergy, uncontrolled thyroid diseases or hypertension, diabetic ketoacidosis, hepatitis B, hepatitis C, HIV.
* Having severe autoimmune/immunodeficiency, macrovascular, renal, or neuromuscular disease, or severe retinopathy or neuropathy.
* Having any other cardiovascular, pulmonary, orthopaedic, neurologic, psychiatric, or terminal disease, or any other acute/chronic disorder that, in the opinion of the local clinician/researcher, would preclude participation and successful completion of the protocol, or that would directly influence the study results.
* Use of any medication (e.g., steroids), that, in the opinion of local clinician/researcher, would negatively impact or mitigate full participation and completion, or could influence the study results.
* Any condition that would interfere with compliance or the results, as judged by the Investigator
* Pregnant women: having multiple pregnancy
* Pregnant women: evidence of incompetent cervix, ruptured membranes, placenta previa, foetal malformation, or foetal death.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in the euglycemic range for the 24 hours after each experimental condition | assessed in the study phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 24 hours/day)
  * T1DM non-pregnant women, euglycemic range: 3.9 - 10 mmol/L (70 - 180 mg/dL).
  * T1DM pregnant women, euglycemic range: 3.5 - 7.8 mmol/L (63 - 140 mg/dL).
Percentage of time spent in the euglycemic range for the 24 hours after each experimental condition | assessed in the study phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 24 h/day)
  * T1DM non-pregnant women: 3.9 - 10 mmol/L (70 - 180 mg/dL).
  * T1DM pregnant women: 3.5 - 7.8 mmol/L (63 - 140 mg/dL).

SECONDARY OUTCOMES:
Percentage of time spent in hypoglycemia for the 24 hours after each experimental condition | assessed in the study phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 24 hours/day)
  * T1DM non-pregnant women - range: < 3.9 mmol/L (< 70 mg/dL).
  * T1DM pregnant women - range: < 3.5 mmol/L (< 63 mg/dL).
Percentage of time spent in hypoglycemia for the 24 hours after each experimental condition | assessed in the study phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 24 h/day)
  * T1DM non-pregnant women - range: < 3.9 mmol/L (< 70 mg/dL).
  * T1DM pregnant women - range: < 3.5 mmol/L (< 63 mg/dL).
Percentage of time spent in hyperglycemia for the 24 hours after each experimental condition | assessed in the study phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 24 hours/day)
  * T1DM non-pregnant women - range: > 10 mmol/L (> 180 mg/dL).
  * T1DM pregnant women - range: > 7.8 mmol/L (> 140 mg/dL).
Percentage of time spent in hyperglycemia for the 24 hours after each experimental condition | assessed in the study phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 24 h/day)
  * T1DM non-pregnant women - range: > 10 mmol/L (> 180 mg/dL).
  * T1DM pregnant women - range: > 7.8 mmol/L (> 140 mg/dL).
Differences in postprandial glucose levels 1-, 2-, and 4-hours post-experiment | assessed in the study phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 4 h/day)
  Within-change in glucose values (mmol/L) from pre-experiment (before starting exercise/meal testing) to post-experiment (i.e., 1-, 2-, and 4-hours after starting exercise/meal intake) in each experimental day
Differences in postprandial glucose levels 1-, 2-, and 4-hours post-experiment | assessed in the study phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 4 h/day)
  Within-change in glucose values (mmol/L) from pre-experiment (before starting exercise/meal testing) to post-experiment (i.e., 1-, 2-, and 4-hours after starting exercise/meal intake) in each experimental day
Number of hypoglycaemic events for the 24 hours after each experimental condition | assessed in the study phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 24 hours/day)
  * T1DM non-pregnant women - range: < 3.9 mmol/L (< 70 mg/dL).
  * T1DM pregnant women - range: < 3.5 mmol/L (< 63 mg/dL).
Number of hypoglycaemic events for the 24 hours after each experimental condition | assessed in the study phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 24 h/day)
  * T1DM non-pregnant women - range: < 3.9 mmol/L (< 70 mg/dL).
  * T1DM pregnant women - range: < 3.5 mmol/L (< 63 mg/dL).
Number of hyperglycaemic events for the 24 hours after each experimental condition | assessed in the study phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 24 hours/day)
  * T1DM non-pregnant women - range: > 10 mmol/L (> 180 mg/dL).
  * T1DM pregnant women - range: > 7.8 mmol/L (> 140 mg/dL).
Number of hyperglycaemic events for the 24 hours after each experimental condition | assessed in the study phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 24 h/day)
  * T1DM non-pregnant women - range: > 10 mmol/L (> 180 mg/dL).
  * T1DM pregnant women - range: > 7.8 mmol/L (> 140 mg/dL).
Percentage of time spent in nocturnal euglycemia within each experimental day | assessed in the study phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 00:00 am - 05:59 am)
  * T1DM non-pregnant women - range: euglycemia 3.9 - 10 mmol/L (70 - 180 mg/dL).
  * T1DM pregnant women - range: euglycaemia 3.5 - 7.8 mmol/L (63 - 140 mg/dL).
Percentage of time spent in nocturnal euglycemia within each experimental day | assessed in the study phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 00:00 am - 05:59 am )
  * T1DM non-pregnant women - range: euglycemia 3.9 - 10 mmol/L (70 - 180 mg/dL).
  * T1DM pregnant women - range: euglycaemia 3.5 - 7.8 mmol/L (63 - 140 mg/dL).
Percentage of time spent in diurnal euglycemia within each experimental day | assessed in the study phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 6.00 am - 23:59 am)
  * T1DM non-pregnant women - range: euglycemia 3.9 - 10 mmol/L (70 - 180 mg/dL).
  * T1DM pregnant women - range: euglycaemia 3.5 - 7.8 mmol/L (63 - 140 mg/dL).
Percentage of time spent in diurnal euglycemia within each experimental day | assessed in the study phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 6.00 am - 23:59 am)
  * T1DM non-pregnant women - range: euglycemia 3.9 - 10 mmol/L (70 - 180 mg/dL).
  * T1DM pregnant women - range: euglycaemia 3.5 - 7.8 mmol/L (63 - 140 mg/dL).
Area under the curve of glycaemic exposure | assessed in the study phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 8 hours/day)
  Area under the curve of glycaemic exposure during the 2, 4 and 8 hours after meal intake at each experimental condition.
Area under the curve of glycaemic exposure | assessed in the study phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 8 h/day)
  Area under the curve of glycaemic exposure during the 2, 4 and 8 hours after meal intake at each experimental condition.
Glycaemic variability (standard deviation) | assessed in the study phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 24 hours/day)
  Standard deviation (SD) of the mean continuous glucose monitoring levels over the 24 hours after each experimental condition
Glycaemic variability (standard deviation) | assessed in the study phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 24 h/day)
  Standard deviation (SD) of the mean continuous glucose monitoring levels over the 24 hours after each experimental condition
Glycaemic variability (coefficient of variation) | assessed in the study phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 24 hours/day)
  Coefficient of variation of glucose levels over the 24 hours after each experimental condition
Glycaemic variability (coefficient of variation) | assessed in the study phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 24 h/day)
  Coefficient of variation of glucose levels over the 24 hours after each experimental condition
Maternal glucose metabolism | assessed in the phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 3 h/day)
  Fasting and post-experiment blood samples will be collected using venous puncture in the antecubital vein. Metabolic markers related to the glucose-insulin axis will be analysed (i.e., glucose, insulin, C-peptide and HbA1c).
Maternal glucose metabolism | assessed in the phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 3 h/day)
  Fasting and post-experiment blood samples will be collected using venous puncture in the antecubital vein. Metabolic markers related to the glucose-insulin axis will be analysed (i.e., glucose, insulin, C-peptide and HbA1c).
Maternal lipid profile | assessed in the phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 3 h/day)
  Fasting and post-experiment blood samples will be collected using venous puncture in the antecubital vein. Metabolic markers related to the lipid profile will be analysed (i.e., total cholesterol, high-density lipoprotein (HDL) cholesterol, LDL-cholesterol, triglycerides and free fatty acids).
Maternal lipid profile | assessed in the phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 3 h/day)
  Fasting and post-experiment blood samples will be collected using venous puncture in the antecubital vein. Metabolic markers related to the lipid profile will be analysed (i.e., total cholesterol, high-density lipoprotein (HDL) cholesterol, LDL-cholesterol, triglycerides and free fatty acids).
Maternal inflammatory markers | assessed in the phase 1 (10 days) - at visit nº 2, 3, 4 (3 days, 3 h/day)
  Fasting and post-experiment blood samples will be collected using venous puncture in the antecubital vein. Metabolic markers related to inflammatory-immunological responses will be analysed (e.g., IL-6, IL-8, IL-1β, TNFα, C-reactive protein, IFNγ)
Maternal inflammatory markers | assessed in the phase 2 (only pregnant women, 10 days) - at visit nº 6, 7, 8 (3 days, 3 h/day)
  Fasting and post-experiment blood samples will be collected using venous puncture in the antecubital vein. Metabolic markers related to inflammatory-immunological responses will be analysed (e.g., IL-6, IL-8, IL-1β, TNFα, C-reactive protein, IFNγ)
Placenta weight | assessed at birth - 30 minutes
  Placenta weight (grams)
Placenta biopsies | collected at birth - 1 hour
  Eight biopsies will be collected, four on the maternal site and four on the fetal side. Relevant placental proteins (growth factors and cytokines) related to insulin signalling, glucose metabolism, and inflammation will be analysed (e.g., GM-CSF, GCSF, MCP1, TNF-α, IL-6, EGF, IFN-γ, IL-8, IL-10, IL-1β).
Neonate weight | assessed at birth - 5 minutes
  Neonate weight (grams)
Placenta efficiency | estimated after birth - 3 minutes
  Neonate weight divided by placenta weight

OTHER OUTCOMES:
Placenta completeness | assessed at birth - 20 minutes
  The number of present and missing cotyledons and velamentous vessels will be examined visually in all the quadrants.
Neonate height | assessed at birth - 5 minutes
  Neonate height (cm)
Neonate ponderal index | estimated after birth - 3 minutes
  Neonate weight/height ratio: 100 x weight / (Height)3
Neonate anthropometrics | assessed at birth - 10 minutes
  Neonate head and abdomen circumference (cm). These circumferences will be measured using a stretch-resistant measuring tape.
Neonate Apgar score | assessed at birth - 5 minutes
  Neonate Apgar score (1-10). The higher score is indicative of a better health status of the newborn after birth
Small for gestational age | assessed after birth - 5 minutes
  Newborns will be diagnosed as small for gestational age newborns if their birth weight is lower than the 10th percentile for their gestational age
Large for gestational age | assessed after birth - 5 minutes
  Newborns will be diagnosed as large for gestational age newborns if their birth weight is greater than the 90th percentile for their gestational age
Physical fitness (muscle strenght) | assessed in the phase 1, at visit nº 1 (10 minutes)
  Upper body muscle strength will be measured by the handgrip strength test.
Physical fitness (muscle strenght) | assessed in the phase 2 (only pregnant women), at visit nº 5 (10 minutes)
  Upper body muscle strength will be measured by the handgrip strength test.
Physical fitness (flexibility) | assessed in the phase 1, at visit nº 1 (10 minutes)
  Upper body flexibility will be assessed by the back scratch test, measuring the distance or overlap between the middle fingers of both hands behind the back.
Physical fitness (flexibility) | assessed in the phase 2 (only pregnant women), at visit nº 5 (10 minutes)
  Upper body flexibility will be assessed by the back scratch test, measuring the distance or overlap between the middle fingers of both hands behind the back.
Physical fitness (cardiorespiratory fitness) | assessed in the phase 1, at visit nº 1 (30 minutes)
  Cardiorespiratory fitness will be assessed using a submaximal walking treadmill test while recording gas exchange data (breath by breath system).
Physical fitness (cardiorespiratory fitness) | assessed in the phase 2 (only pregnant women), at visit nº 5 (30 minutes)
  Cardiorespiratory fitness will be assessed using a submaximal walking treadmill test while recording gas exchange data (breath by breath system).
Resting energy expenditure | assessed in the phase 1, at visit nº 1 (2 hours)
  Gas exchange will be measured breath by breath using a portable gas analyser
Physical activity | assessed in the phase 1 - 10 continuous days
  Physical activity levels will be measured with triaxial accelerometry.
Physical activity | assessed in the phase 2 (only pregnant women) - 10 continuous days
  Physical activity levels will be measured with triaxial accelerometry.
Vital signs (systolic and diastolic blood pressure) | assessed in the phase 1, at visit nº 1 (15 minutes)
  Systolic and diastolic blood pressure (mmHg) will be assessed twice using an upper arm digital sphygmomanometer with women seated, relaxed and not talking.
Vital signs (systolic and diastolic blood pressure) | assessed in the phase 2 (only pregnant women), at visit nº 5 (15 minutes)
  Systolic and diastolic blood pressure (mmHg) will be assessed twice using an upper arm digital sphygmomanometer with women seated, relaxed and not talking.
Vital signs (resting heart rate) | assessed in the phase 1, at visit nº 1 (15 minutes)
  Resting heart rate (beats per minute) will be assessed twice using an upper arm digital sphygmomanometer with women seated, relaxed and not talking.
Vital signs (resting heart rate) | assessed in the phase 2 (only pregnant women), at visit nº 5 (15 minutes)
  Resting heart rate (beats per minute) will be assessed twice using an upper arm digital sphygmomanometer with women seated, relaxed and not talking.
Initial anamnesis (sociodemographic and clinical information) | assessed in the phase 1, at visit nº 1 (40 minutes)
  Relevant information from the patients will be collected by the physicians who will ask them, and by an initial questionnaire prepared by the researchers (e.g., age, educational level, occupational status, medications, diseases, etc.).
Sleep quality (questionnaire) | assessed in the phase 1, at visit nº 1 (20 minutes)
  The sleep quality will be assessed using a validated questionnaire, the Pittsburgh Sleep Quality Index questionnaire (PSQI). Higher scores indicate worse sleep quality (0-21).
Sleep quality (questionnaire) | assessed in the phase 2 (only pregnant women), at visit nº 5 (20minutes)
  The sleep quality will be assessed using a validated questionnaire, the Pittsburgh Sleep Quality Index questionnaire (PSQI). Higher scores indicate worse sleep quality (0-21).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Acosta-Manzano, PhD, Principal Investigator — University of Graz; Mireille van Poppel, Principal Investigator — University of Graz
Locations (1):
- University of Graz, Graz, Styria, Austria